CLINICAL TRIAL: NCT07180667
Title: Acute Effects of Different Warm-Up Protocols on Motor Performance in Adolescent Football Goalkeepers: A Randomised Crossover Study
Brief Title: Warm-Up Effects on Adolescent Goalkeepers' Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, bekir tokay, Instructor of Physical Education and Sport, Faculty of Sport Sciences, Ph.D., Uşak University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 207-01-08; Uşak University (Other: 207-01-08)
Record Dates: First submitted 2025-09-02; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Healhty; Adolescent; Football; Warm-up
Keywords: Warm-up protocols,; Youth goalkeepers; Motor performance; Dynamic stretching; Balance; Explosive strength
MeSH Terms: interventions — Warm-Up Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: No additional parties are masked in this study. Only the outcome assessors are blinded to the warm-up protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Aerobic Running Warm-Up (AR) (Experimental): Participants perform a 15-minute aerobic running protocol with heart rate maintained at 60-75% of age-predicted maximum (HRₘₐₓ). Includes 7 minutes of light jogging followed by slight intensity increase.
  Interventions: Behavioral: Intervention 1: Aerobic Running (AR) Warm-Up
- Arm 2: Static Stretching Warm-Up (SS) (Experimental): Participants perform 5 minutes of light jogging, followed by static stretches of six lower-limb muscle groups (gastrocnemius, quadriceps, hamstrings, hip flexors, adductors, gluteals). Each muscle stretched twice for 30 seconds. Finishes with 3-4 minutes of light dynamic movements.
  Interventions: Behavioral: Intervention 2: Static Stretching (SS) Warm-Up
- Arm 3: Dynamic Stretching Warm-Up (DS) (Experimental): Participants perform 5 minutes of light jogging, followed by dynamic stretches targeting the same six lower-limb muscle groups over 10-15 meters with short rest between repetitions.
  Interventions: Behavioral: Intervention 3: Dynamic Stretching (DS) Warm-Up
- Arm 4: Movement Preparation Warm-Up (MP) (Experimental): Participants perform a combination of light jogging, multi-joint mobility drills (e.g., lateral shuffles, inchworms), submaximal sprinting (80-90% maximum velocity), and low-intensity balance drills adapted from FIFA 11+ and HarmoKnee.
  Interventions: Behavioral: Intervention 4: Movement Preparation (MP) Warm-Up

INTERVENTIONS:
Behavioral: Intervention 1: Aerobic Running (AR) Warm-Up — 15-minute aerobic running protocol. Heart rate maintained at 60-75% of age-predicted maximum (HRₘₐₓ). Includes 7 minutes light jogging followed by slight intensity increase.
  Arms: Arm 1: Aerobic Running Warm-Up (AR)
Behavioral: Intervention 2: Static Stretching (SS) Warm-Up — 5 minutes light jogging followed by static stretches of six lower-limb muscles (gastrocnemius, quadriceps, hamstrings, hip flexors, adductors, gluteals). Each muscle stretched twice for 30 seconds, finishing with 3-4 minutes of light dynamic movements.
  Arms: Arm 2: Static Stretching Warm-Up (SS)
Behavioral: Intervention 3: Dynamic Stretching (DS) Warm-Up — 5 minutes light jogging followed by dynamic stretches targeting the same six muscle groups over 10-15 meters with brief rest between repetitions.
  Arms: Arm 3: Dynamic Stretching Warm-Up (DS)
Behavioral: Intervention 4: Movement Preparation (MP) Warm-Up — Description: Combination of light jogging, multi-joint mobility drills (e.g., lateral shuffles, inchworms), submaximal sprinting (80-90% max velocity), and low-intensity balance drills adapted from FIFA 11+ and HarmoKnee.
  Arms: Arm 4: Movement Preparation Warm-Up (MP)

SUMMARY:
The purpose of this study is to examine the acute effects of different warm-up protocols on performance outcomes in adolescent male football goalkeepers. Specifically, it investigates the impact of aerobic running, static stretching, dynamic stretching, and movement preparation on flexibility, explosive power, and dynamic balance.

DETAILED DESCRIPTION:
This randomized crossover study examined the acute effects of four 15-minute warm-up protocols-Aerobic Running (AR), Static Stretching (SS), Dynamic Stretching (DS), and Movement Preparation (MP)-on flexibility, explosive lower-limb power, and dynamic balance in 15 adolescent male football goalkeepers. Participants were licensed youth goalkeepers with consistent sleep, diet, and training routines. Warm-up order was randomized and both participants and administrators were blinded to the condition. Flexibility, power, and balance were assessed using the sit-and-reach test, standing long jump, and Y Balance Test, respectively, with the best of three trials recorded. Heart rate was monitored to maintain internal load at 60-75% of age-predicted maximum. All sessions were supervised by a certified sports scientist, and anthropometric data were collected prior to testing. Ethical approval and informed consent were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Biologically male football goalkeepers
* Aged 14-15 years
* Actively competing in youth leagues
* Minimum training experience of approximately 3-4 years
* Free from chronic diseases or musculoskeletal injuries that could affect physical performance
* Maintain regular sleep and dietary routines during the study period

Exclusion Criteria:

* Current injuries
* Chronic health conditions
* Any physical limitations that could interfere with safe participation in warm-up protocols or performance testing

Ages: 14 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Only male participants are eligible.
Enrollment: 15 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Flexibility (Sit and Reach) | Immediately post-intervention, after each warm-up session (4 sessions, separated by at least 48 hours).
  Flexibility of the posterior chain was assessed using the sit-and-reach test with a standardized measurement box. Participants performed three trials barefoot with knees fully extended, and the best score was recorded in centimeters.
Explosive Lower-Limb Power (Standing Long Jump) | Immediately post-intervention, after each warm-up session (4 sessions, separated by at least 48 hours).
  Explosive horizontal power was measured by the standing long jump test. From a standing position, participants jumped bilaterally as far as possible. The distance was measured to the nearest cm from the starting line to the rearmost heel. Three maximal trials were performed with 2 minutes rest, and the best score was used.
Dynamic Balance (Y Balance Test normalized composite score) | Immediately post-intervention, after each warm-up session (4 sessions, separated by at least 48 hours).
  Dynamic postural control was assessed using the Y Balance Test. Reach distances in the anterior, posteromedial, and posterolateral directions were normalized to leg length. A composite score (mean of three directions) was calculated and used for analysis.

SECONDARY OUTCOMES:
Anthropometric Parameters (Height, Weight, BMI) | Baseline (Day 1, prior to the first warm-up intervention session)
  Body height (cm), body weight (kg), and BMI (kg/m²) measured with stadiometer and electronic scale prior to warm-up interventions.
Internal Load (Heart Rate Monitoring) | During each warm-up session (15 minutes, across AR, SS, DS, MP protocols)
  Heart rate continuously monitored with Polar RS300X. Intensity calibrated to maintain 60-75% of age-predicted HRmax, calculated individually using Tanaka formula [208 - (0.7 × age)].

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa AKIL, Professor Dr., Principal Investigator — Uşak University; Melek G. GUNGOR, Principal Investigator — Uşak University; Mehmet Emin Yelken, Ph.D., Principal Investigator — Ilgaz Provincial Directorate of Youth and Sports
Locations (1):
- Uşak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
A definitive plan regarding the sharing of individual participant data has not been established at this time